CLINICAL TRIAL: NCT03248271
Title: Effects of Insulin on Hypotension and Sarcopenia
Status: Withdrawn | Type: Observational
Why Stopped: Study design was changed to the study was changed to Insulin, hypotension and sarcopenia.
Sponsor: Kenneth Madden (Other)
Responsible Party: Sponsor-Investigator, Kenneth Madden, Associate Professor, UBC Department of Medicine, University of British Columbia
Organization: University of British Columbia (Other)
Other Study IDs: H17-01663
Record Dates: First submitted 2017-08-07; First posted 2017-08-14 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Diabetes; Sarcopenia; Hypotension, Orthostatic
Keywords: Diabetes; Sarcopenia; Hypotension; Tilt Table Test
MeSH Terms: conditions — Diabetes Mellitus; Sarcopenia; Hypotension, Orthostatic; Hypotension | interventions — Insulin Lispro

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetes, Insulin Naive: Study participants will be tested prior to and 3 and 6 months after starting insulin to manage their diabetes
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Lispro — Insulin
  Other Names: Humalog

SUMMARY:
In this study investigator's aim to determine the impact of insulin therapy on hypotension and sarcopenia

DETAILED DESCRIPTION:
Diabetes is common in the elderly. By the age of 70, approximately 25% of the population has diabetes and another 25% is at risk for diabetes. Elderly patients with diabetes are at increased risk for disability and reduction in their instrumental and basic activities of daily living. The prevalence of frailty is higher in people with diabetes that with age matched controls without diabetes. One of the major contributing factors to frailty is sarcopenia.

Insulin is an important anabolic hormone that prevents protein breakdown and to a lesser extent stimulates protein synthesis. There is some evidence that the ability of insulin to stimulate anabolic processes may be reduced in diabetes.

Insulin has cardiovascular properties, resulting in simultaneous adrenergic and vasodilatory responses that have opposing influences on blood pressure. Epidemiological studies have demonstrated that the use of insulin is a risk factor for syncope.

The investigators will study 30 older adults age 65 and older with type 2 diabetes who have never taken insulin to manage their diabetes but now need insulin to manage their diabetes. Data will be compared pre insulin start and 3 and 6 months after starting insulin.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Type 2 diabetes for at least 5 years
* Insulin naive
* now needs insulin to manage diabetes

Exclusion Criteria:

* anemia as defined by serum hematocrit
* abnormal liver function tests
* elevated serum creatinine
* smoked within last 5 years
* musculoskeletal or neurological condition that would preclude tilt table testing or orthostatic vitals
* aortic stenosis

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Older adults age 65 and older with type 2 diabetes who do not use insulin to manage their diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Body composition | Change from months 0, 3 and 6 months post insulin start
  Measured by DEXA Scan
Grip strength | Change from months 0, 3 and 6 months post insulin start
  measured by Hand Dynamometer
Physical functioning Survey | Change from months 0, 3 and 6 months post insulin start
  measured by the Physical Component Summary from the SF-12 Health
Presence or absence of orthostatic hypotension | Change from months 0, 3 and 6 months post insulin start
  Drop in systolic blood pressure of greater than 20 mmHg after 3 minutes of standing
Nadir of systolic blood pressure during the Tilt Table Test | Change from months 0, 3 and 6 months post insulin start
  Lowest systolic blood pressure obtained during the Tilt Table Test
Nadir of diastolic blood pressure during the Tilt Table Test | Change from months 0, 3 and 6 months post insulin start
  Lowest diastolic blood pressure obtained during the Tilt Table Test

SECONDARY OUTCOMES:
Nadir of middle cerebral artery velocity as measured by transcranial doppler | Change from months 0, 3 and 6 months post insulin start
  Lowest middle cerebral artery velocity obtained during the Tilt Table Test
Presence or absence of a positive Tilt Table Test (vasovagal syncope) | Change from months 0, 3 and 6 months post insulin start
  Sudden drop in blood pressure and heart rate that leads to fainting

CONTACTS AND LOCATIONS:
Overall Officials: Madden M Kenneth, MD, Principal Investigator — University of British Columbia/Gerontology Research Lab
Locations (1):
- University of British Columbia - Gerontology Research Lab, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morley JE, Malmstrom TK, Rodriguez-Manas L, Sinclair AJ. Frailty, sarcopenia and diabetes. J Am Med Dir Assoc. 2014 Dec;15(12):853-9. doi: 10.1016/j.jamda.2014.10.001. Epub 2014 Nov 20. No abstract available. PMID 25455530
- [Background] Rizzo MR, Barbieri M, Fava I, Desiderio M, Coppola C, Marfella R, Paolisso G. Sarcopenia in Elderly Diabetic Patients: Role of Dipeptidyl Peptidase 4 Inhibitors. J Am Med Dir Assoc. 2016 Oct 1;17(10):896-901. doi: 10.1016/j.jamda.2016.04.016. Epub 2016 Jun 2. PMID 27262494
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Meneilly GS, Knip A, Tessier D. Diabetes in the elderly. Can J Diabetes. 2013 Apr;37 Suppl 1:S184-90. doi: 10.1016/j.jcjd.2013.01.045. Epub 2013 Mar 26. No abstract available. PMID 24070944
- [Background] Leenders M, Verdijk LB, van der Hoeven L, Adam JJ, van Kranenburg J, Nilwik R, van Loon LJ. Patients with type 2 diabetes show a greater decline in muscle mass, muscle strength, and functional capacity with aging. J Am Med Dir Assoc. 2013 Aug;14(8):585-92. doi: 10.1016/j.jamda.2013.02.006. Epub 2013 Mar 26. PMID 23537893
- [Background] Bassil MS, Gougeon R. Muscle protein anabolism in type 2 diabetes. Curr Opin Clin Nutr Metab Care. 2013 Jan;16(1):83-8. doi: 10.1097/MCO.0b013e32835a88ee. PMID 23196814
- [Background] Salle A, Guilloteau G, Ryan M, Bouhanick B, Ritz P. Effect of insulin treatment on the body composition of Type 2 diabetic patients. Diabet Med. 2004 Dec;21(12):1298-303. doi: 10.1111/j.1464-5491.2004.01335.x. PMID 15569132
- [Background] Gin H, Rigalleau V, Perlemoine C. Insulin therapy and body weight, body composition and muscular strength in patients with type 2 diabetes mellitus. J Nutr Metab. 2010;2010:340570. doi: 10.1155/2010/340570. Epub 2009 Oct 21. PMID 20721344
- [Background] de Kanter M, Lilja B, Elmstahl S, Eriksson KF, Sundkvist G. A prospective study of orthostatic blood pressure in diabetic patients. Clin Auton Res. 1998 Aug;8(4):189-93. doi: 10.1007/BF02267780. PMID 9791738
- [Background] Gupta V, Lipsitz LA. Orthostatic hypotension in the elderly: diagnosis and treatment. Am J Med. 2007 Oct;120(10):841-7. doi: 10.1016/j.amjmed.2007.02.023. PMID 17904451
- [Background] Vinik AI, Erbas T. Cardiovascular autonomic neuropathy: diagnosis and management. Curr Diab Rep. 2006 Dec;6(6):424-30. doi: 10.1007/s11892-006-0074-z. PMID 17118224
- [Background] Tack CJ, Lenders JW, Willemsen JJ, van Druten JA, Thien T, Lutterman JA, Smits P. Insulin stimulates epinephrine release under euglycemic conditions in humans. Metabolism. 1998 Mar;47(3):243-9. doi: 10.1016/s0026-0495(98)90251-7. PMID 9500557
- [Background] Tack CJ, Smits P, Willemsen JJ, Lenders JW, Thien T, Lutterman JA. Effects of insulin on vascular tone and sympathetic nervous system in NIDDM. Diabetes. 1996 Jan;45(1):15-22. doi: 10.2337/diab.45.1.15. PMID 8522054
- [Background] Meneilly GS, Elliott T, Battistini B, Floras JS. N(G)-monomethyl-L-arginine alters insulin-mediated calf blood flow but not glucose disposal in the elderly. Metabolism. 2001 Mar;50(3):306-10. doi: 10.1053/meta.2001.19493. PMID 11230783
- [Background] Lipsitz LA, Pluchino FC, Wei JY, Rowe JW. Syncope in institutionalized elderly: the impact of multiple pathological conditions and situational stress. J Chronic Dis. 1986;39(8):619-30. doi: 10.1016/0021-9681(86)90187-6. PMID 3090090
- [Background] Ruiz GA, Calvar C, Hermes R, Rivadeneira D, Bengolea V, Chirife R, Tentori MC, Gelpi RJ. Insulin sensitivity in young women with vasovagal syncope. Am Heart J. 2003 May;145(5):834-40. doi: 10.1016/S0002-8703(02)94707-1. PMID 12766740
- [Background] Stratton JR, Cerqueira MD, Schwartz RS, Levy WC, Veith RC, Kahn SE, Abrass IB. Differences in cardiovascular responses to isoproterenol in relation to age and exercise training in healthy men. Circulation. 1992 Aug;86(2):504-12. doi: 10.1161/01.cir.86.2.504. PMID 1638718
- [Background] Madden KM, Tedder G, Lockhart C, Meneilly GS. Euglycemic hyperinsulinemia alters the response to orthostatic stress in older adults with type 2 diabetes. Diabetes Care. 2008 Nov;31(11):2203-8. doi: 10.2337/dc08-1058. Epub 2008 Aug 20. PMID 18716048
- [Background] Sergi G, De Rui M, Stubbs B, Veronese N, Manzato E. Measurement of lean body mass using bioelectrical impedance analysis: a consideration of the pros and cons. Aging Clin Exp Res. 2017 Aug;29(4):591-597. doi: 10.1007/s40520-016-0622-6. Epub 2016 Aug 27. PMID 27568020
- [Background] Ziegler D, Laux G, Dannehl K, Spuler M, Muhlen H, Mayer P, Gries FA. Assessment of cardiovascular autonomic function: age-related normal ranges and reproducibility of spectral analysis, vector analysis, and standard tests of heart rate variation and blood pressure responses. Diabet Med. 1992 Mar;9(2):166-75. doi: 10.1111/j.1464-5491.1992.tb01754.x. PMID 1563252
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Del Rosso A, Ungar A, Bartoli P, Cellai T, Mussi C, Marchionni N, Masotti G; Gruppo Italiano di Studio Della Sincope Dell'anziano. Usefulness and safety of shortened head-up tilt testing potentiated with sublingual glyceryl trinitrate in older patients with recurrent unexplained syncope. J Am Geriatr Soc. 2002 Aug;50(8):1324-8. doi: 10.1046/j.1532-5415.2002.50351.x. PMID 12164986
- [Background] Lipsitz LA, Mukai S, Hamner J, Gagnon M, Babikian V. Dynamic regulation of middle cerebral artery blood flow velocity in aging and hypertension. Stroke. 2000 Aug;31(8):1897-903. doi: 10.1161/01.str.31.8.1897. PMID 10926954